CLINICAL TRIAL: NCT00683592
Title: A Randomized, Double-blind, Placebo Controlled Study Assessing the Efficacy and Safety of Vilazodone 40 mg qd and Evaluating Genetic Biomarkers Associated With Treatment Response in Patients With Major Depressive Disorder (MDD)
Brief Title: Randomized, Double-Blind, Placebo Controlled Study of Vilazodone's Efficacy, Safety, and Biomarkers of Response in Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Carol R. Reed, MD, PGxHealth, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDA-07-DP-02
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): vilazodone
  Interventions: Drug: vilazodone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vilazodone — titration to 40 mg tablets qd (once a day) for 8 weeks
  Other Names: EMD68843, SB-659746
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter, 8-week, clinical trial is designed to assess the efficacy and safety of vilazodone and to evaluate genetic biomarkers of treatment response associated with vilazodone use in adult patients diagnosed with MDD by the DSM-IV-TR criteria.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multicenter, 8-week, clinical trial is designed to assess the efficacy and safety of vilazodone and to evaluate genetic biomarkers of treatment response associated with vilazodone use in adult patients diagnosed with MDD by the DSM-IV-TR criteria. This study will enroll approximately 470 patients at approximately 10 clinical sites. Safety and efficacy will be assessed at each visit. A DNA sample will be collected and analyzed for response to vilazodone.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years of age.
* A diagnosis of MDD, single episode or recurrent, according to DSM-IV-TR (296.2/296.3) with a current Major Depressive Episode of less than two year's duration with a minimum duration of at least 4 weeks.
* Meets DSM-IV-TR criteria for Major Depressive Disorder.
* HAM-D score ≥ 22 on the first 17 items of the 21-item HAM-D.
* HAM-D item 1 (depressed mood) score ≥ 2.
* Patients must be able to provide written informed consent
* Patients must be able to speak, read and understand English

Exclusion Criteria:

* Patients with a current (or within 6 months prior to the Screening Visit) Axis I disorder of Post Traumatic Stress Disorder, Eating Disorder, Obsessive Compulsive Disorder.
* Patients with a history of schizophrenia, schizoaffective disorder or bipolar I or II disorder (with a history of hypomanic or manic episodes).
* Patients who meet DSM-IV-TR criteria for substance abuse (alcohol or drugs) within 3 months prior to the Screening Visit or substance dependence within 6 months prior to the Screening Visit.
* Patients who meet criteria for any of the following DSM-IV-TR MDD Specifiers: [a] With Catatonic Features; [b] With Postpartum Onset; [c] With Seasonal Pattern [d]severe with Psychotic Features.
* Patients who are receiving formal psychotherapy or have had psychotherapy within the 12 weeks prior to the Screening Visit.
* Patients who have any one of the following:

  * In the month prior to screening, have had active suicidal ideation with some intent to act, without specific plan.
  * In the month prior to screening, have had suicidal ideation with specific plan and intent.
  * Have made a suicide attempt within the 6 months prior to the screening visit.
  * In the opinion of the Investigator, is currently at significant risk of suicide.
* Patients who have had an inadequate response to at least 2 consecutive antidepressants from different classes given at adequate doses for an adequate duration.
* Patients who have received electroconvulsive therapy within the 6 months prior to the Screening Visit.
* Patients currently taking a psychotropic drug. Patients who have taken psychotropic drugs must have discontinued these prior to the Screening Visit. The minimum discontinuation periods are outlined in the study protocol.
* Patients taking migraine medications with a serotonergic mechanism of action
* Patients taking CYP3A4 inhibitors such as grapefruit juice, ketoconazole, diltiazem, and macrolide antibiotics or montelukast
* Patients with known hypersensitivity to SSRIs (selective serotonin reyptake inhibitors) or 5-HT1a agonists.
* Patients previously treated with vilazodone (also known as SB-659746-A or EMD 68 843).
* Patients with a history of clinically significant cardiac, renal, neurologic, cerebrovascular, hepatic, hematologic, metabolic or pulmonary disorders.
* Patients with any serious medical disorder or condition that would, in the investigator's opinion, preclude the administration of study medication.
* Female patients must not be pregnant, lactating, or planning to become pregnant during the time of study participation. All female patients must be at least 1 year post menopausal or irreversibly surgically sterilized (by hysterectomy, oophorectomy, or bilateral tubal ligation with resection) or determined not to be at risk of pregnancy.
* Patients with clinically significant abnormalities on electrocardiogram.
* Patients having clinically significant abnormal laboratory findings.
* Patients with a positive drug screen.
* Patients who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures.
* Patients that have taken an investigational drug or participated in an investigational drug trial within the past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol R Reed, MD, Study Director — Forest Laboratories
Locations (9):
- United States (9):
  - Pharmacology Research Institute, Newport Beach, California
  - Florida Clinical Research Center, Bradenton, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Summit Research Network, Portland, Oregon
  - University of Pennsylvania Department of Psychiatry Mood and Anxiety Disorders, Philadelphia, Pennsylvania
  - Mood Disorders Research Program and Clinic Exchange Park, Dallas, Texas
  - University of Utah Health Sciences Ctr, Dept of Psychiatry Mood Disorders Clinic, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network, Seattle, Washington

REFERENCES:
- [Derived] Kornstein S, Chang CT, Gommoll CP, Edwards J. Vilazodone efficacy in subgroups of patients with major depressive disorder: a post-hoc analysis of four randomized, double-blind, placebo-controlled trials. Int Clin Psychopharmacol. 2018 Jul;33(4):217-223. doi: 10.1097/YIC.0000000000000217. PMID 29608461
- [Derived] Culpepper L, Mathews M, Ghori R, Edwards J. Clinical relevance of vilazodone treatment in patients with major depressive disorder: categorical improvement in symptoms. Prim Care Companion CNS Disord. 2014;16(1):PCC.13m01571. doi: 10.4088/PCC.13m01571. Epub 2014 Jan 30. PMID 24940525
- [Derived] Jain R, Chen D, Edwards J, Mathews M. Early and sustained improvement with vilazodone in adult patients with major depressive disorder: post hoc analyses of two phase III trials. Curr Med Res Opin. 2014 Feb;30(2):263-70. doi: 10.1185/03007995.2013.855188. Epub 2013 Oct 31. PMID 24127687
- [Derived] Clayton AH, Kennedy SH, Edwards JB, Gallipoli S, Reed CR. The effect of vilazodone on sexual function during the treatment of major depressive disorder. J Sex Med. 2013 Oct;10(10):2465-76. doi: 10.1111/jsm.12004. Epub 2012 Dec 6. PMID 23216998
- [Derived] Reed CR, Kajdasz DK, Whalen H, Athanasiou MC, Gallipoli S, Thase ME. The efficacy profile of vilazodone, a novel antidepressant for the treatment of major depressive disorder. Curr Med Res Opin. 2012 Jan;28(1):27-39. doi: 10.1185/03007995.2011.628303. Epub 2011 Nov 23. PMID 22106941
- [Derived] Khan A, Cutler AJ, Kajdasz DK, Gallipoli S, Athanasiou M, Robinson DS, Whalen H, Reed CR. A randomized, double-blind, placebo-controlled, 8-week study of vilazodone, a serotonergic agent for the treatment of major depressive disorder. J Clin Psychiatry. 2011 Apr;72(4):441-7. doi: 10.4088/JCP.10m06596. PMID 21527122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was 31Mar2008 to 10Feb2009.
Pre-assignment Details: This study included a washout period to allow patients to discontinue their current antidepressant medications and any additional medications prohibited by the protocol, if applicable.
Groups:
- Vilazodone: Vilazodone titrated to 40mg. Two tablets per day.
- Placebo: Placebo to match vilazodone. Two tablets per day.
Period: Overall Study
Arm/Group | Vilazodone | Placebo
Started | 240 | 241
Intent to Treat Population | 231 | 232
Safety Population | 235 | 233
Completed | 193 | 195
Not Completed | 47 | 46
Not completed — Adverse Event | 12 | 4
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 17 | 17
Not completed — Lack of Efficacy | 3 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Non-compliance | 3 | 5
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vilazodone (ITT Population): Vilazodone, 40 mg
- Placebo (ITT Population): placebo to match vilazodone
- Total: Total of all reporting groups
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population) | Total
Number analyzed (Participants) | 231 | 232 | 463
Age Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.22) | 42.4 (12.49) | 41.7 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 123 | 261
  Male | 93 | 109 | 202
Region of Enrollment [Number; unit: participants]
  United States | 231 | 232 | 463

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the MADRS (Montgomery-Asberg Depression Rating Scale) Total Score.
Description: The MADRS is an observer rating scale that has proven to be an efficient and practical measure of depression. The scale was constructed to be sensitive to treatment effects. The change from baseline in MADRS total score has a possible range of -60 to 60 where negative values reflect improvement in depression symptom severity. The method of last observation carried forward was utilized for subjects who discontinued prematurely.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Week 8
Population: Intent-to-Treat (ITT): the ITT population consisted of patients who were randomized, took at least 1 dose of study drug, and had at least 1 post-baseline efficacy endpoint measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Units on a scale | -13.3 [-15.1 to -11.5] | -10.8 [-12.6 to -9.1]
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); The model was an analysis of covariance (ANCOVA), with terms for treatment group and center, adjusting for baseline MADRS total score. Missing values at week 8 were handled using the last observation carried forward (LOCF) approach; Test type: Superiority or Other; p = 0.009, ANCOVA; Difference in Least Squares Mean Change = -2.5, 95% CI 2-sided [-4.4 to -0.6]

2. Secondary Outcome: Change From Baseline to Week 8 in the HAM-D 17 (17-Item Hamilton Rating Scale for Depression) Total Score
Description: The HAM-D 17 is a 17-item subscale of the HAM-D 21, which is designed to be completed by a trained rater. It is designed for rating depressive symptom severity in patients with a confirmed diagnosis of depressive disorder. The change in HAM-D 17 has a possible range of -52 to 52 with negative values indicating improvment in depression symptom severity. The method of last observation carried forward was utilized for subjects who discontinued prematurely.
Time Frame: Baseline, week 1, week 2, week 4, week 6, week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Units on a scale | -10.7 [-12.1 to -9.4] | -9.1 [-10.4 to -7.7]
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); The model was an analysis of covariance (ANCOVA), with terms for treatment group and center, adjusting for baseline HAM-D 17 total score. Missing values at week 8 were handled using the last observation carried forward (LOCF) approach; Test type: Superiority or Other; p = 0.026, ANCOVA; Difference in Least Squares Mean Change = -1.6, 95% CI 2-sided [-3.1 to -0.2]

3. Secondary Outcome: The CGI-I (Clinician's Global Impression of Improvement) Score at Week 8
Description: The CGI-I scale measures change from the baseline state at every visit after the baseline visit. It permits a global evaluation of the patient's improvement over time. At the scheduled clinic visits, the clinician assessed the patient's improvement relative to the symptoms at baseline on a CGI-I item using a 7-point scale, where 1 = very much improved and 7 = very much worse. The method of last observation carried forward was utilized for subjects who discontinued prematurely.
Time Frame: Week 1, Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Units on a scale | 2.5 [2.3 to 2.7] | 2.8 [2.6 to 3.0]
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); The model was an analysis of variance (ANOVA), with terms for treatment group and center. Missing values at week 8 were handled using the last observation carried forward (LOCF) approach; Test type: Superiority or Other; p = 0.004, ANOVA; Difference in Least Squares Mean Improve = -0.3, 95% CI 2-sided [-0.5 to -0.1]

4. Secondary Outcome: Change From Baseline to Week 8 in the HAM-A ( Hamilton Anxiety Rating Scale) Total Score
Description: The HAM-A is a rating scale developed to quantify the severity of anxiety. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe). Change from baseline in the HAM-A total score may range from -52 to 52 with negative value indicating improvement in anxiety symptom severity. The method of last observation carried forward was utilized for subjects who discontinued prematurely.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Units on a scale | -7.0 [-8.0 to -5.9] | -5.7 [-6.8 to -4.7]
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); The model was an analysis of covariance (ANCOVA), with terms for treatment group and center, adjusting for baseline HAM-A total score. Missing values at week 8 were handled using the last observation carried forward (LOCF) approach; Test type: Superiority or Other; p = 0.037, ANCOVA; Difference in Least Squares Mean Change = -1.2, 95% CI 2-sided [-2.4 to -0.1]

5. Secondary Outcome: MADRS (Montgomery-Asberg Depression Rating Scale) Response Rate at Week 8
Description: MADRS response was defined as ≥ 50% decrease from baseline in MADRS total score at Week 8. The response rate is the percentage of subjects in each treatment group meeting the criteria for response. The method of last observation carrier forward was utilized for subjects who discontinued prematurely.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Participants | 101 | 70
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); Cochran-Mantel-Haenszel tests were used to compare MADRS response rates between the treatment groups, stratifying by center. The asymptotic confidence interval of the risk difference was estimated by the normal approximation to the binomial distribution; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.134, 95% CI 2-sided [0.047 to 0.221]

6. Secondary Outcome: MADRS (Montgomery-Asberg Depression Rating Scale) Remission Rate at Week 8
Description: MADRS remission was defined as a MADRS total score < 10 at Week 8. The remission rate is the percentage of subjects in each treatment group who met the criteria for remission. The method of last observation carried forward was utilized for subjects who discontinued prematurely.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Vilazodone (ITT Population) | Placebo (ITT Population)
Number analyzed (Participants) | 231 | 231
Participants | 63 | 47
Statistical Analysis 1: Comparison: Vilazodone (ITT Population) vs Placebo (ITT Population); Cochran-Mantel-Haenszel tests were used to compare MADRS remission rates between the treatment groups, stratifying by center. The asymptotic confidence interval of the risk difference was estimated by the normal approximation to the binomial distribution; Test type: Superiority or Other; p = 0.066, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.069, 95% CI 2-sided [-0.008 to 0.147]

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Vilazodone (Safety Population): Vilazodone, 40mg
- Placebo (Safety Population): placebo to match vilazodone
Arm/Group | Vilazodone (Safety Population) | Placebo (Safety Population)
Serious Adverse Events (participants affected / at risk) | 4/235 | 2/233
Other Adverse Events (participants affected / at risk) | 148/235 | 85/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilazodone (Safety Population) (N=235) | Placebo (Safety Population) (N=233)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) — This subject also had the SAE of carotid arteriosclerosis.
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) — This subject also had the SAE of angina pectoris
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilazodone (Safety Population) (N=235) | Placebo (Safety Population) (N=233)
Abnormal Dreams (Psychiatric disorders) | 14 (14) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 72 (91) | 25 (35)
Dizziness (Nervous system disorders) | 21 (21) | 9 (9)
Dry Mouth (Gastrointestinal disorders) | 21 (21) | 9 (10)
Headache (Nervous system disorders) | 30 (32) | 24 (25)
Insomnia (Psychiatric disorders) | 17 (22) | 7 (7)
Nausea (Gastrointestinal disorders) | 61 (71) | 13 (15)
Upper Respiratory Infections (Infections and infestations) | 8 (8) | 21 (21)
Vomiting (Gastrointestinal disorders) | 12 (13) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators have the right to publish or permit the publication of any information or material relating to or arising out of this protocol after prior submission to PGxHealth provided that, if PGxHealth requests, the investigator will delay publication for a maximum of six months to enable PGxHealth to protect their rights in such information or material.